CLINICAL TRIAL: NCT02278185
Title: An Open Label, Randomized, Phase II Trial of Metabolic Complications in Patients Treated With Enzalutamide vs Standard ADT for the Treatment of Hormone Sensitive Prostate Cancer
Brief Title: Enzalutamide Versus Standard Androgen Deprivation Therapy for the Treatment Hormone Sensitive Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-0909.cc; NCI-2014-02219 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Results first posted 2022-04-27 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Leuprolide; Goserelin; histrelin; Triptorelin Pamoate; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (enzalutamide) (Experimental): Patients receive enzalutamide PO QD for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enzalutamide
- Arm II (ADT) (Active Comparator): Patients receive standard of care ADT comprising one of the following at the discretion of the treating physician: leuprolide acetate, goserelin acetate, histrelin acetate, triptorelin, or degarelix SC or IM for 12 months in the absence of disease progression or unacceptable toxicity. Patients may also choose to undergo surgical castration as an alternative form of ADT.
  Interventions: Drug: leuprolide acetate; Drug: goserelin acetate; Drug: histrelin acetate; Drug: triptorelin; Drug: degarelix

INTERVENTIONS:
Drug: Enzalutamide — Given PO
  Other Names: MDV3100; selective androgen receptor modulator MDV3100; XTANDI
  Arms: Arm I (enzalutamide)
Drug: leuprolide acetate — Given SC or IM
  Other Names: Enantone; LEUP; Lupron; Lupron Depot
  Arms: Arm II (ADT)
Drug: goserelin acetate — Given SC or IM
  Other Names: ICI-118630; ZDX; Zoladex
  Arms: Arm II (ADT)
Drug: histrelin acetate — Given SC or IM
  Other Names: Supprelin; Vantas
  Arms: Arm II (ADT)
Drug: triptorelin — Given SC or IM
  Other Names: 6-D-Tryptophan-LH-RH; 6-D-Tryptophanluteinizing Hormone-releasing Factor; D-TRP-6-LHRH; Decapeptyl; TRIP
  Arms: Arm II (ADT)
Drug: degarelix — Given SC or IM
  Other Names: ASP3550; FE200486; Firmagon
  Arms: Arm II (ADT)

SUMMARY:
This randomized phase II trial compares enzalutamide with standard androgen deprivation therapy in reducing incidence of metabolic syndrome in patients with prostate cancer that has spread to other places in the body. Metabolic syndrome is defined as changes in cholesterol, blood pressure, circulating sugar levels, and body weight. Previous studies have shown that patients with prostate cancer, who have been treated with standard medical therapy that lowers testosterone levels, have an increased risk of these changes. Hormone therapy using enzalutamide may fight prostate cancer by blocking the use of testosterone by the tumor cells instead of lowering testosterone levels. It is not yet known whether prostate cancer patients who receive enzalutamide will have reduced incidence of metabolic syndrome than patients who receive standard androgen deprivation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the incidence of metabolic syndrome within 12 months, as defined by the Adult Treatment Panel III, in patients treated with enzalutamide compared to standard androgen deprivation therapy.

SECONDARY OBJECTIVES:

I. To determine the incidence of metabolic syndrome within 6 months, as defined by the Adult Treatment Panel III, in patients treated with enzalutamide compared to standard androgen deprivation therapy.

II. To assess bone health, as measured by a dual-energy x-ray absorptiometry (DXA) scanner.

III. To assess body composition (sarcopenic obesity), as measured by a DXA scanner.

IV. To assess quality of life (QOL), as measured by the Functional Assessment of Cancer Therapy-Prostate (FACT-P) and Sexual Health Inventory in Men (SHIM).

V. To assess time to prostate-specific antigen (PSA) progression and time to radiographic progression.

VI. To assess the incidence of developing individual risk factors, or components, which comprise metabolic syndrome.

VII. To assess the change in high-sensitivity C-reactive protein (hs-CRP) as a marker of inflammation.

VIII. To assess the safety and tolerance of enzalutamide or androgen deprivation therapy (ADT).

IX. To assess the change in physical function as measured by the Short Physical Performance Battery (SPPB).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive enzalutamide orally (PO) once daily (QD) for 12 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive standard of care ADT comprising one of the following at the discretion of the treating physician: leuprolide acetate, goserelin acetate, histrelin acetate, triptorelin, or degarelix subcutaneously (SC) or intramuscularly (IM) for 12 months in the absence of disease progression or unacceptable toxicity. Patients may also choose to undergo surgical castration as an alternative form of ADT.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the prostate; if pathology is unavailable, the principal investigator (PI) may also make a determination of prostate cancer based on unequivocal clinic data
* Patients with advanced prostate cancer suitable for systemic treatment defined as: having metastatic disease, a biochemical relapse after primary therapy, or patients in whom primary therapy is not appropriate or feasible; patients without metastatic disease will need evaluation for local therapy and deemed inappropriate or have refused this treatment option
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Age > 18 years
* Must use a condom if having sex with a pregnant woman
* A male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration
* Life expectancy estimated at > 12 months
* Ability to understand and willingness to provide written informed consent document

Exclusion Criteria:

* A history of androgen deprivation therapy; patients receiving hormonal therapy in the adjuvant and/or neoadjuvant setting must have discontinued therapy at least 6 months prior to day 1 of treatment AND have a serum testosterone level >= 50 ng/dL AND cannot have received more than 18 months of previous ADT
* A history of orchiectomy
* Previous androgen blockade (e.g. antiandrogens) in the last 3 months
* Patients already meeting the criteria for metabolic syndrome as defined by the Adult Treatment Panel III Criteria which requires 3/5 parameters encompassing glucose control, blood pressure, lipids and waist circumference; patients with 2 of the parameters at baseline will be allowed enrollment provided that one of those risk factors is hypertension (>= 130/>= 85 mm Hg)
* Baseline hypogonadism as defined as a testosterone < 50 ng/dL
* PSA < 0.5 ng/dL
* Serum vitamin D 25, hydroxy (OH) < 12 ng/mL
* Active hepatitis C virus
* Use of corticosteroids as defined by a daily dose of prednisone (or equivalent) of 5 mg or greater for more than 1 month continuously within 3 months of screening
* Corrected calcium > 10.6 mg/dL
* Absolute neutrophil count < 1500/uL
* Platelet count < 100,000/uL
* Hemoglobin < 9 g/dL
* Total bilirubin >= 1.5 x upper limit of normal (ULN) (unless documented Gilbert's)
* Alanine aminotransferase or aspartate aminotransferase >= 2.5 x ULN
* Creatinine > 2 mg/dL
* Clinically significant cardiovascular disease as evidenced by: myocardial infarction within 6 months of screening; uncontrolled angina within 3 months of screening; New York Heart Association (NYHA) class 3 or 4 congestive heart failure; clinically significant ventricular arrhythmia; Mobitz II/2nd degree/or 3rd degree heart block without a pacemaker in place; uncontrolled hypertension (HTN) (systolic > 180 mmHg or diastolic > 105 mmHg at screening)
* Previous exposure to enzalutamide
* Use of an investigational therapeutic within 30 days
* History of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study agent
* Known or suspected brain metastasis or active leptomeningeal disease
* History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke, significant brain trauma) at any time in the past; also, history of loss of consciousness or transient ischemic attack within 12 months of day 1 visit
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2024-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Kessler, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Health - Poudre Valley Hospital, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
Started | 10 | 9
Completed | 7 | 7
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT) | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Median (Full Range); unit: years] | 62 [56 to 77] | 68 [56 to 86] | 66 [56 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
PSA value [Median (Full Range); unit: NG/ML] | 10.86 [2.1 to 105.97] | 5.48 [0.87 to 23.7] | 7.55 [0.87 to 105.97]
Metastatic disease [Count of Participants; unit: Participants] | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Syndrome Incidence, Summarized by the Number of Patients With at Least 3 of the 5 Pre-specified Criteria
Description: Metabolic syndrome will be assessed at the beginning of each course and defined by the presence of 3 of the following five traits: abdominal obesity, defined as a waist circumference > 102 cm (> 40 in); serum triglycerides >= 150 mg/dL (1.7 mmol/L) or drug treatment for elevated triglycerides; serum high density lipoprotein (HDL) cholesterol < 40 mg/dL (1 mmol/L) or drug treatment for low HDL; blood pressure >= 130/>= 85 mmHg or drug treatment for elevated blood pressure; and fasting plasma glucose (FPG) >= 100 mg/dL (5.6 mmol/L) or drug treatment for elevated blood glucose.
Time Frame: Within the first 12 months of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
Number analyzed (Participants) | 10 | 9
Participants | 5 | 3
Statistical Analysis 1: Comparison: Arm I (Enzalutamide) vs Arm II (ADT); The difference between metabolic syndrome and treatment were evaluated with the Chi-square test; Test type: Superiority; p = 0.46, Chi-squared; This study did not meet it's target accrual goal and thus is underpowered to detect a statistically significant difference between the two groups
Statistical Analysis 2: Comparison: Arm I (Enzalutamide) vs Arm II (ADT); Cohort characteristics for Metabolic Syndrome were summarized by event and arm using counts and percentages for categorical variables and the mean, standard deviation, median, and quartiles for continuous variables. The difference between metabolic syndrome and treatment were evaluated with the Chi-square test. P-values are reported based on a null hypothesis of no difference against a two-sided alternative. Analyses were performed using SAS 9.4 (SAS Inst; Test type: Superiority; p = 0.46, Chi-squared; Cohort characteristics for Metabolic Syndrome, the SPPB, the SHIM/FACT-P, and PSA were summarized by event and arm using counts and percentages for categorical variables and the mean, standard deviation, median, and quartiles for continuous variables. The difference between metabolic syndrome and treatment were evaluated with the Chi-square test. The Wilcoxon signed-rank test was utilized to examine the difference between Month 1 and Month 12 SPPB scores. The Wilcoxon rank-sum test was used to assess the difference of SHIM/FACT-P scores and PSA between arms. These tests were chosen to account for the non-normal distributions of the continuous variables. The difference between PSA progression between arms was examined using the Fisher Exact Test. A heat map of scores ordered by the highest average score was also created. P-values are reported based on a null hypothesis of no difference against a two-sided alternative. Analyses were performed using SAS 9.4 (SAS Inst

2. Secondary Outcome: Metabolic Syndrome Incidence, Summarized by the Proportion of Patients With at Least 3 of the 5 Pre-specified Criteria
Description: Metabolic syndrome will be assessed at the beginning of each course and defined by the presence of 3 of the following five traits: abdominal obesity, defined as a waist circumference > 102 cm (> 40 in); serum triglycerides >= 150 mg/dL (1.7 mmol/L) or drug treatment for elevated triglycerides; serum HDL cholesterol < 40 mg/dL (1 mmol/L) or drug treatment for low HDL; blood pressure >= 130/>= 85 mmHg or drug treatment for elevated blood pressure; and FPG >= 100 mg/dL (5.6 mmol/L) or drug treatment for elevated blood glucose.
Time Frame: Within the first 6 months of therapy
Population: Includes all patients still participating at this timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
Number analyzed (Participants) | 10 | 9
Participants | 4 | 0

3. Secondary Outcome: Change in Bone Turnover Markers, as Measured by Bone-specific Alkaline Phosphatase
Description: Will be assessed for each treatment group. Measurements will be taken at day 1 of each course. A paired t-test will test within an arm as to whether the change from baseline to 12 months is significantly different from zero.
Time Frame: Baseline and month 12
Population: Patients were compared to themselves as well as across groups. We reviewed difference from month 1 to 12 in order to gather adequate data. Below are the bone-specific alkaline phosphatase. Not all patients completed follow up for this measure.
Measure: Mean (Standard Deviation); unit: microgram/L
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
Number analyzed (Participants) | 4 | 5
microgram/L | -18.55 (36.19) | -58.14 (133.53)

4. Secondary Outcome: Change in Bone Density
Description: We will measure bone density via a DXA scanner, Left Femur and Right femur T scores will be added to a composite score. A paired t-test will test within an arm as to whether the change from baseline to twelve months is significantly different from zero.
  The T-score is the standard deviation of how much bone density differs from the bone mass of an average healthy 30 year old. A score of 0 indicates no deviation from average. The following ranges are used:
  * T-score of -1.0 or above = normal bone density
  * T-score between -1.0 and -2.5 = low bone density, or osteopenia
  * T-score of -2.5 or lower = osteoporosis
Time Frame: Baseline to 12 months
Population: Not all patients completed follow-up for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Enzalutamide: Patients exposed to enzalutamide
- Androgen Deprivation Therapy: Patients exposed to androgen deprivation therapy
Arm/Group | Enzalutamide | Androgen Deprivation Therapy
Number analyzed (Participants) | 4 | 5
score on a scale | -0.23 (0.26) | 0 (0.29)

5. Secondary Outcome: Change in Free Fat Mass, as Measured by a DXA Scanner
Description: A paired t-test will test within an arm as to whether the change from baseline to each time point is significantly different from zero.
  These data are not able to be reported as the DXA did not measure free fat mass and thus we will be using cross sectional CT analysis.
Time Frame: Baseline to up to 12 months
Population: The DXA scanner was not able to analyze free fat mass, only bone density.
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Fat Mass, as Measured by a DXA Scanner
Description: A paired t-test will test within an arm as to whether the change from baseline to each time point is significantly different from zero.
Time Frame: Baseline to up to 12 months
Population: data cannot be reported as the dexa scanner used for the study only measured bone density and not lean body mass (this was realized part way through study).
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Quality of Life (QOL) Scores, as Measured by the Functional Assessment of Cancer Therapy - Prostate (FACT-P) and Sexual Health in Men (SHIM)
Description: The FACT-P is the Functional Assessment of Cancer Therapy - Prostate and measures physical/emotional quality of life in prostate cancer patients.
  NUMBER OF ITEMS:39 PATIENT POPULATION:Prostate cancer patients 18 years and older RECALL PERIOD:Past 7 days RESPONSE SCALE:5 point Likert-type scale
  SUBSCALE DOMAINS:
  Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), Functional Well-Being (FWB), Prostate Cancer Subscale (PCS)
  SCORING:
  Scores range from 0-158. In general, the higher the score, the better the quality of life.
  Sexual Health in Men (SHIM). 5 item measure of erectile function. Total score is 1-25 with a higher score indicating better sexual health. Scores: no ED (SHIM total score, 22-25), mild (17-21), mild to moderate (12-16), moderate (8-11), and severe ED (1-7).
Time Frame: Baseline to up to 7 months
Population: Patients were compared to themselves as well as across groups. We reviewed difference from month 1 to 7 in order to gather adequate data. Below is the SHIM.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
Number analyzed (Participants) | 10 | 9
score on a scale
  SHIM: number analyzed (Participants) | 7 | 5
  SHIM | -3.71 (5.06) | -3.4 (5.98)
  FACT-P: number analyzed (Participants) | 8 | 5
  FACT-P | -4.5 (10.15) | -1.93 (6.82)

8. Secondary Outcome: Number of Patients With PSA Progression
Description: PSA progression as defined by an increase in >= 50% from nadir and an absolute increase of at least 2 ng/mL above the nadir, occurring at least 12 weeks after start of therapy that is confirmed by two consecutive increases taken at least 2 weeks apart. Log rank test will be used to compare the distributions of above variables between the group treated with enzalutamide to the group on standard ADT.
Time Frame: Time from randomization to the earliest objective evidence of PSA progression as defined per protocol, assessed up to 30 days after the last dose of study drug
Population: All patients were evaluated throughout the course of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
Number analyzed (Participants) | 10 | 9
Participants | 0 | 1

9. Secondary Outcome: Time to Radiographic Progression
Description: Log rank test will be used to compare the distributions of above variables between the group treated with enzalutamide to the group on standard ADT.
Time Frame: Time from randomization to the earliest objective evidence of radiographic progression as defined per protocol, assessed up to 30 days after the last dose of study drug
Population: All participants included in analysis.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
Number analyzed (Participants) | 10 | 9
Months | NA (NA) — No patients on study experienced radiographic progression within the study period. | 11.474 (NA) — Only one patient experienced radiographic progression within the study period.

10. Secondary Outcome: Change in Markers of Inflammation, as Measured by Circulating Hs-CRP
Description: Mean change in available samples from baseline to 12 months, presented in mg/dL
Time Frame: Difference between baseline and 12 months.
Population: Patients were compared to themselves as well as across groups. We reviewed difference from month 1 to 12 in order to gather adequate data. Some patients in the cohort were missing follow-up data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
Number analyzed (Participants) | 6 | 6
mg/dL | 0.87 (1.99) | 6.42 (16.47)

11. Secondary Outcome: Incidence of Adverse Events, Using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.1
Description: The incidence of adverse events has been reported in the adverse events log for clinicaltrials.gov
Time Frame: Up to 30 days after the last dose of study drug
Population: adverse events reported in separate section
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide | Androgen Deprivation Therapy
Number analyzed (Participants) | 10 | 9
Participants | 10 | 9

12. Secondary Outcome: Change in Physical Function, as Measured by Short Physical Performance Battery (SPPB).
Description: The Short SPPB incorporates 3 validated portions to assess a patient's balance and mobility. SPPB scores range from zero to 12 possible points. SPPB score of 3-9 points in persons with no mobility disability indicates frailty; SPPB score of 10 or greater for persons with no sarcopenia and no mobility disability indicates robustness. The higher the score, the better the physical function. Will be measured as a continuous outcome.
Time Frame: Difference between baseline and 12 months.
Population: Not all patients completed follow-up for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
Number analyzed (Participants) | 5 | 6
score on a scale | 10.58 (1.39) | 10.94 (1.97)
Statistical Analysis 1: Comparison: Arm I (Enzalutamide) vs Arm II (ADT); The results are presented in the following format: N Mean (Std Dev) Median (Q1, Q3). In all cases (Overall, Arm 1, and Arm 2) we fail to reject the null hypothesis that the samples come from the same population of scores at Month 1 versus Month 12 at the 0.05 significance level; Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Change in Bone Turnover Markers as Measured by N-telopeptide
Description: Will be assessed for each treatment group. Measurements will be taken at day 1 of each course. A paired t-test within an arm as to whether the change from baseline to 12 months is significantly different from zero. N-Telopeptide units - nM Bone Collagen Equivalent (BCE).
Time Frame: Baseline and 12 months
Population: Patients were compared to themselves as well as across groups. We reviewed difference from month 1 to 12 to gather adequate data. Below are the N-telopeptide. Not all patients completed follow-up for this measure.
Measure: Mean (Standard Deviation); unit: nM BCE
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
Number analyzed (Participants) | 6 | 7
nM BCE | -3.05 (5.51) | 1.73 (8.41)

ADVERSE EVENTS:
Time Frame: Monitoring of adverse events was conducted throughout the study. These were reported from the date written informed consent and through 30 days post-last dose of study drug.
Description: There is no difference in our definition of an adverse event and that of clinicaltrials.gov
Arm/Group | Arm I (Enzalutamide) | Arm II (ADT)
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/9
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/9
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Enzalutamide) (N=10) | Arm II (ADT) (N=9)
Subarachnoid Hemmorhage (Nervous system disorders) | 0 (0) | 1 (1)
Radiation esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 4 elevation in triglycerides possibly related to study treatment and resolved in folow up.
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Enzalutamide) (N=10) | Arm II (ADT) (N=9)
abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
activity change (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
alcohol abuse (Social circumstances) | 0 (0) | 2 (2)
Allergic rhinitis (Immune system disorders) | 1 (1) | 0 (0)
ALT increase (Hepatobiliary disorders) | 0 (0) | 3 (3)
anal bleeding (Gastrointestinal disorders) | 0 (0) | 3 (3)
anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
arthralgias (Immune system disorders) | 7 (7) | 8 (8)
ast increase (Hepatobiliary disorders) | 1 (1) | 2 (2)
ataxia (Nervous system disorders) | 0 (0) | 1 (1)
back pain (General disorders) | 6 (6) | 4 (4)
Basal cell skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
jaw pain (General disorders) | 1 (1) | 0 (0)
hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 1 (1) | 1 (1)
cognitive changes (Nervous system disorders) | 2 (2) | 0 (0)
Constipation (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Dark urine (Renal and urinary disorders) | 1 (1) | 0 (0)
Decreased concentration (Nervous system disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dizziness (General disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ear other (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Elevated triglyceride (Cardiac disorders) | 2 (2) | 0 (0)
erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Eye disorders (other) (Eye disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (6) | 5 (5)
flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 10 (11) | 2 (2)
Alopecia (Immune system disorders) | 1 (1) | 1 (1)
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hep A (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hot Flashes (General disorders) | 3 (3) | 9 (9)
hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Endocrine disorders) | 1 (1) | 1 (1)
vision change (Eye disorders) | 0 (0) | 1 (1)
insomnia (General disorders) | 1 (1) | 3 (3)
cough (General disorders) | 2 (2) | 0 (0)
nasal congestion (Immune system disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Loose stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
memory change (Psychiatric disorders) | 1 (1) | 0 (0)
myalgias (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Rhinorrhea (Immune system disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 1 (1) | 4 (4)
Neck pain (General disorders) | 1 (1) | 2 (2)
creatnine increased (Renal and urinary disorders) | 0 (0) | 1 (1)
decreased libido (Reproductive system and breast disorders) | 0 (0) | 1 (1)
neuropathy (Nervous system disorders) | 1 (1) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Movements involuntary (Nervous system disorders) | 1 (1) | 0 (0)
middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
radiculitis (Nervous system disorders) | 1 (1) | 1 (1)
dehydration (General disorders) | 0 (0) | 1 (1)
sinus congestion (Immune system disorders) | 1 (1) | 2 (2)
Sleep disturbance (General disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
dental problems (General disorders) | 0 (0) | 1 (1)
tinnitus (Ear and labyrinth disorders) | 1 (1) | 3 (3)
dysguesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
tremors (Nervous system disorders) | 1 (1) | 0 (0)
Weight gain (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
emotional lability (Psychiatric disorders) | 0 (0) | 1 (1)
Voice alteration (General disorders) | 1 (1) | 0 (0)
weakness (General disorders) | 1 (1) | 3 (3)
Weight loss (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
epistaxis (Ear and labyrinth disorders) | 0 (0) | 2 (2)
esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
facial swelling (General disorders) | 0 (0) | 1 (1)
fall (General disorders) | 0 (0) | 1 (1)
hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)
nystagmus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
influenza (General disorders) | 0 (0) | 1 (1)
seizure (Nervous system disorders) | 0 (0) | 1 (1)
edema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
lymphocyte decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
night sweats (Nervous system disorders) | 0 (0) | 1 (1)
injection site reaction (Surgical and medical procedures) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Sneezing (Immune system disorders) | 0 (0) | 1 (1)
spinal cord compression (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
subarachnoid hemmorhage (Nervous system disorders) | 0 (0) | 1 (1)
trouble swallowing (Nervous system disorders) | 0 (0) | 1 (1)
urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was originally designed when ADT alone was SOC treatment for metastatic prostate cancer. In the years of opening and enrollment, the SOC changed thus affecting the population of potentially eligible patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT02278185/Prot_SAP_000.pdf